CLINICAL TRIAL: NCT03185936
Title: Pars Plana Vitrectomy With Internal Limiting Membrane Peeling in Optic Disc Pit Maculopathy
Brief Title: Surgical Management of Optic Disc Pit Maculaopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mahmoud Genaidy, Assistant professor of ophthalmology, Minia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ODP-M
Record Dates: First submitted 2017-06-09; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Optic Disc Structural Anomaly; Maculopathy
Keywords: optic disc pit; retinal detachment; maculopathy
MeSH Terms: conditions — Macular Degeneration; Retinal Detachment | interventions — Tooth Exfoliation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Optic disc pit maculopathy (Experimental): pars plana vitrectomy with internal limiting membrane (ILM) peeling, endolaser
  Interventions: Procedure: pars plana vitrectomy with internal limiting membrane (ILM) peeling

INTERVENTIONS:
Procedure: pars plana vitrectomy with internal limiting membrane (ILM) peeling — pars plana vitrectomy (PPV) combined with internal limiting membrane (ILM) peeling, endolaser photocoagulation and gas tamponade in management of optic disc pit (ODP) maculopathy.
  Other Names: Endolaser photocoagulation

SUMMARY:
To evaluate the anatomical and functional results of pars plana vitrectomy (PPV) combined with internal limiting membrane (ILM) peeling, endolaser photocoagulation and gas tamponade in management of optic disc pit (ODP) maculopathy.

DETAILED DESCRIPTION:
As it is well known, optic disc pit (ODP) is a rare congenital disease which is usually associated with maculopathy (ODP-M) in the form of intraretinal and subretinal fluid accumulation at the macular area leading to visual impairment.

With no definite treatment and absence of guidelines for its management, the invistigators considered their prospective, interventional case series to evaluate the anatomical and functional results of pars plana vitrectomy (PPV) combined with internal limiting membrane (ILM) peeling, endolaser photocoagulation and gas tamponade in management of optic disc pit (ODP) maculopathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in this study are those with ODP associated with macular detachment

Exclusion Criteria:

* Exclusion criteria included patients unfit for general anesthesia, those with insufficient clear media to perform the surgery with ILM peeling and those with other ocular diseases that can affect central macular thickness (CMT) and the best corrected visual acuity (BCVA).

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-03-01 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
anatomical improvement | 6 months
  Retinal reattachment

SECONDARY OUTCOMES:
Functional improvement | 6 months
  Visual acuity letters gain

CONTACTS AND LOCATIONS:
Overall Officials: Mahmud Genaidy, MD, Principal Investigator — Assistant professor of ophthalmology, ophthalmology department, Minia university, Egypt

IPD SHARING:
Plan to Share IPD: No
Can not be shared